CLINICAL TRIAL: NCT01013493
Title: Association Between Breastfeeding and Likelihood of Myopia in 6-7 Years Old Children
Status: Completed | Type: Observational
Sponsor: National Nutrition and Food Technology Institute (Other)
Responsible Party: Amin Salehi Abargouei, SBMU, National Nutrition and Food Technology Research Institute (NNFTRI)
Other Study IDs: 292
Record Dates: First submitted 2009-11-12; First posted 2009-11-13 (Estimated); Last update posted 2009-12-02 (Estimated); Status verified 2009-12

CONDITIONS: Myopia; Nearsightedness
Keywords: breastfeeding; myopia; nearsightedness; children
MeSH Terms: conditions — Myopia; Breast Feeding

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- myopic
- non myope-healthy

SUMMARY:
Myopia is the main reason of vision loss in the world which is seen in 30.4 million adults in USA (1). In a myopic eye, images are focused in front of retina because, cornea and crystalline lens become more powerful in focusing the image or the eye axis become too long (axial myopia) (2).

Myopia prevalence in adolescents has been raised in recent years and nowadays it has reached to 10-25% and 60-80% in western and eastern countries respectively (3). Tehran eye study showed that the prevalence of myopia in Tehran is 21.8% and 17.2% based on manifest and cycloplegic refraction respectively (4). One study in Dezful, Iran showed that 3.7% of 7-15 years old children are myopic (5).

Today potential role of early life nutrition in myopia development in later life is becoming an attractive field of study. It has been shown that until weaning; breast milk is the main source of many nutrients [such as docosahexaenoic acid (DHA)] which are important for photoreceptors and cortical neuronal development (6). But results about the relationship between breastfeeding and likelihood of childhood myopia are controversial. A hypothesis-generating study (7) showed an independent and inverse relationship between breastfeeding and likelihood of myopia in 10-12 year old Singaporean children. However, data pulled from three English birth cohorts done in 10-11y and 15-16y children did not show any effect (8).

To examine the association between breastfeeding pattern and likelihood of myopia in 6-7y children, a retrospective case-control study is designed in National Nutrition and Food Technology research Institute of Iran. This study will try to assess breastfeeding pattern and almost all cofactors which may relate to myopia.

DETAILED DESCRIPTION:
For proper vision, eyes need to focus exactly on images. The two main determinants of refraction are focus power of cornea and the eye's axis length. In normal eyes, images are formed exactly on retina (emmetropia), but farsightedness (hyperopia) is the situation in which, the eye forms images in the backside of retina and nearsightedness (myopia) is a situation in which images are formed in front of retina, and it may have two reasons: 1) the lens convexity is more powerful than normal and 2) the eye axis is longer than normal (axial myopia).

Refractive errors are measured in diopter (D), and myopia is specified with a negative sign. Severity of myopia is categorized into 3 levels. 1) Mild (0 to -1.5D), 2) moderate (-1.5D to -6.0D) and 3) and severe myopia (-6.0D or above). Pathogenic myopia develops, when this condition advances to -8.0 D and above. Visual disorders - moderate retina disorders, cataract, and glaucoma - may be seen in patients with moderate and severe myopia. At birth, most infants are hyperopic but this condition lowers when they grow up and by the age 5-8, eyes must be emmetropic (normal and without any refractive error) (2).

Nearsightedness is seen in 30.4 million adults in USA (1). It's prevalence in adolescents is remarkably increased in last decades and today its prevalence in industrialized western and eastern societies are increased into 10-25 and 60-80 percent respectively (3). For American society, 60 percent of myopia can be categorized as early myopia (in childhood/school ages) which is usually in ages 9-11 years, and increases in adolescence years, and decreases in late adolescence and beginning of 20th decade of life, and usually stops at -3 to -4 D(9,10). A study in Tehran (4) showed that prevalence of myopia is 21.8 and 56.6 percent based on manifest and cycloplegic refraction respectively. Another study showed a high prevalence of myopia in schoolchildren from Kashan, Iran (11). Also a study in Dezful, Iran showed that prevalence of myopia in 7-15y and 14-18y children are 3.4 and 33 percent respectively (12).

Factors related to myopia can be divided into two groups: 1) hereditary and 2) environmental. Relationship between heredity and likelihood of myopia has been shown in many studies (13, 14). These studies obviously showed the effect of parental myopia on moderate levels of childhood myopia. Today different areas on several chromosomes are known for severe myopia (such like 18p, 12q, 7q36, TGIF) (15-17). Although it seems that two of these chromosomes (18q, 12q) do not have any relationship with childhood myopia (18).

Environmental factors which studies have shown that may be in relation with myopia are: near work (19, 20), stature (21, 22), night time light exposure (10) [however this relationship was not confirmed neither in American (20) and English children and nor in Indian monkeys (23, 24)], day time light exposure (25), refined sugar consumption [It has been shown that carbohydrate consumption can stimulate a series of events which lead to eye's axial length increase and consequently myopia. So refined sugar consumption which has been increased nowadays may play a role.] (26), IQ (Intelligence quotient) (27-33), birth weight, social and economic condition (7), physical activity (32), and breastfeeding (7).

Increasing prevalence of myopia, particularly in Asian urban children, confirms that life style in childhood and infancy may play a role (3). Today potential effect of early life nutrition on myopia development in later life is becoming an attractive field of study. Breastfeeding has been related to neural development which affects visual acuity. Up to weaning, breastfeeding is the main source of many micronutrients [including docosahexanoic acid (DHA)], which are important for light receptors and brain neural development (6). A study which was done in Singapore showed that breastfeeding is independently related to likelihood of myopia after controlling for cofactors (7). But this study had some limitations which may affect the results. This study had a small population size and its participants were from one school. All factors relating to myopia were not controlled by this study. However, data pulled from three English birth cohorts done in 10-11y and 15-16y children did not show any effect (8). Hence, results about the relationship between breastfeeding and likelihood of childhood myopia are controversial.

To examine the association between breastfeeding pattern and likelihood of myopia in 6-7y children, a retrospective case-control study is designed in National Nutrition and Food Technology research Institute of Iran. This study will try to assess almost all cofactors which may relate to myopia; such as child's age, sex, height, birth weight, maternal age at delivery, IQ (intelligence quotient), near work, parental education and ethnicity, parental myopia, child n-3(omega-3) fatty acid and refined carbohydrate intake, maternal n-3 fatty acid intake, n-3 fatty acid intake while infancy, physical activity and other confounding factors which may have an effect on the relationship among breastfeeding pattern and myopia.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for case group subjects:

* Subjects must be 6-7 years old
* Subjects must have myopia with or without astigmatism and the time period between diagnosis of myopia and recruiting the subjects must not be more than 6 months.
* Subject must be graduating in grade 1 in one of north Tehran elementary schools.
* Subject and their parents must have tendency to participate in this study.

Inclusion criteria for control group subjects:

* Subjects must be 6-7 years old
* Subjects must graduate in grade, class and elementary school which case subjects is graduating in.

Exclusion Criteria:

Exclusion criteria for case group subjects:

* Subjects must not have any eye disorder other than myopia with or without astigmatism
* Subjects must not have any metabolic or congenital disorder which has relationship with myopia.

Exclusion criteria for control group subjects:

* Subjects must not have any eye disorder
* Subjects must not have any metabolic or congenital disorder which has relationship with myopia.
* Subjects must not go on diet for any reason.

Ages: 6 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: This study is a retrospective case-control trial, in which subjects for case and control groups will be chosen based on inclusion and exclusion criteria, from 6-7 years old school children living in north Tehran.
Sampling Method: Non-Probability Sample
Enrollment: 245 (Actual)
Dates: Start 2008-09; Primary Completion 2009-03 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amin Salehi Abargouei, M.S, Principal Investigator — Faculty of Nutrition Sciences and Food Technology, Sh. Beheshti University of Medical Sciences and Health Services, Tehran, Iran; Naser Kalantari, Pediatrist, Study Chair — Faculty of Nutrition Sciences and Food Technology, Sh. Beheshti University of Medical Sciences and Health Services, Tehran, Iran
Locations (1):
- National Nutrition and Food Technology Research Institute (NNFTRI), Tehran, Tehran Province, Iran